CLINICAL TRIAL: NCT06954363
Title: Effectiveness of Muscle Energy Techniques and Mulligan Mobilization Along With Conventional Physical Therapy in Knee Joint Osteoarthritis Patients: A Randomized Controlled Trial
Brief Title: Effectiveness of Muscle Energy Techniques and Mulligan Mobilization Along With Conventional Physical Therapy in Knee Joint Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMU/DIR/CTU/2024/015
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Muscle Stretching Exercises; Range of Motion, Articular
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel treatment groups that includes experimental Group (Mulligan Mobilization + Conventional Physical Therapy) and Control Group (Muscle Energy Technique + Conventional Physical Therapy).
Who Masked: Participant
Masking Description: The study will utilize a single-blinded design, where the patients will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive Mulligan Mobilization combined with Conventional Physical Therapy. Mulligan Mobilization includes medial and lateral tibial glides using a Mulligan belt. Each session will consist of 3 sets of 10 repetitions, administered 5 days a week for 3 weeks. In addition, patients will undergo standard conventional physical therapy exercises such as quadriceps strengthening, straight leg raising, and stretching exercises. Each treatment session will last 30 minutes.
  Interventions: Procedure: Mulligan Mobilization
- Control Group (Active Comparator): Participants in this group will receive Muscle Energy Technique (MET) targeting the hamstring muscles, in combination with Conventional Physical Therapy. The MET will follow a post-isometric relaxation approach, using both direct and indirect methods depending on patient condition. Each isometric contraction will be held for 10 seconds, followed by a 20-second stretch, repeated for 3 sets. Therapy will be conducted 5 days a week over a 3-week period. Each session will last 30 minutes. The same conventional physical therapy regimen as the intervention group will be applied.
  Interventions: Procedure: Muscle Energy Technique (MET)

INTERVENTIONS:
Procedure: Mulligan Mobilization — Mulligan Mobilization involves manual tibial glides (medial and lateral) using a mobilization belt. The patient lies supine with the knee flexed between 30°-45°. The therapist applies a sustained glide while the patient actively moves the knee into flexion and extension. The treatment is delivered in 3 sets of 10 repetitions per session, 5 days per week for 3 weeks, along with a conventional physical therapy protocol.
  Arms: Intervention Group
Procedure: Muscle Energy Technique (MET) — Muscle Energy Technique involves the application of post-isometric relaxation targeting hamstring muscles. The therapist applies a 10-second isometric contraction at the resistance barrier, followed by a 20-second passive stretch, progressing into a new range of motion. This technique is applied 3 times per session, 5 days per week for 3 weeks, in combination with a conventional physical therapy protocol.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the effectiveness of integrating Muscle Energy Technique (MET) and Mulligan Mobilization with conventional physical therapy in the management of knee osteoarthritis (OA), with a specific focus on improving hamstring flexibility and reducing functional limitations. The findings will help inform clinical decision-making and enhance patient outcomes in OA rehabilitation.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive degenerative joint disease characterized by the destruction of articular cartilage and the formation of bone spurs, leading to pain, joint stiffness, and decreased functional mobility. While its exact cause remains unknown, factors such as age, sex, obesity, sedentary lifestyle, genetics, bone density, smoking, and joint location contribute significantly to its development. As patients experience pain and reduced joint mobility, they often limit movement, particularly of the knee, resulting in muscular tightness-most notably in the hamstring, a two-joint muscle.

Globally, OA is a major public health concern, with knee OA affecting approximately 250 million people in 2010, including 18% of women and 9.6% of men over 60. It has substantial economic impacts, such as costing the United States 1-2.5% of its GDP and Spain €4.7 billion in 2007. Regional data from South Asia show higher prevalence in rural populations, emphasizing the disease's widespread burden.

Physical therapy has been shown to be highly effective in managing knee OA symptoms. Several randomized controlled trials support the use of techniques like Muscle Energy Technique (MET) and Mulligan Mobilization. MET has demonstrated superior efficacy compared to static stretching and whole-body vibration in improving hamstring flexibility and reducing stiffness. Similarly, Mulligan Mobilization, particularly when combined with supervised exercises, has shown better outcomes than Maitland mobilization in improving flexibility and function in OA patients.

However, current literature presents conflicting evidence regarding the individual efficacy of MET and Mulligan Mobilization. This study seeks to address these inconsistencies by investigating the effectiveness of integrating both MET and Mulligan Mobilization with conventional physical therapy in treating knee OA. The goal is to provide evidence-based insights that can guide clinicians in optimizing therapeutic strategies for better functional outcomes and enhanced quality of life for patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of osteoarthritis (Grade 1 to 3)
* X-ray showing Grades I to III on Kellgren Lawrence scale of Osteoarthritis.
* Residents of Peshawar verified via NADRA CNIC
* Both genders will be included with unilateral or bilateral knee involvement.
* Age group 40 and above.
* Duration of Knee pain for more than 3 months.

Exclusion Criteria:

* History of any previously known neurological conditions i.e. stroke, peripheral neuropathy
* Fractures in treatment limb.
* Suspicious of malignancy around the knee joint.
* Recent under gone surgery
* Recent Intra-articular injection.
* Significant comorbid diseases and disabilities are excluded from the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Hamstring Flexibility Measured by Goniometer | Baseline (Day 1) and Post-treatment (End of Week 3)
  Hamstring range of motion (ROM) will be assessed using a goniometer before and after the intervention. The change in ROM will be used to evaluate effectiveness. Outcome improvement categories:
  Mild Increase: 5-10 degrees
  Moderate Increase: 10-15 degrees
  Marked Increase: >15 degrees
Change in Pain Score Using Knee Osteoarthritis Outcome Score-12 questionnaire Questionnaire | Baseline (Day 1) and Post-treatment (End of Week 3)
  The function in daily activities subscale of Knee Osteoarthritis Outcome Score-12 questionnaire will assess participants' ability to perform routine activities before and after the intervention.
Change in Knee-Related Quality of Life Using Knee Osteoarthritis Outcome Score-12 questionnaire | Baseline (Day 1) and Post-treatment (End of Week 3)
  The quality of life (QOL) subscale of KOOS-12 will evaluate the impact of osteoarthritis on participants' knee-related wellbeing pre- and post-treatment.
Change in Activity of Daily Living Function Using KOOS-12 | Baseline (Day 1) and Post-treatment (End of Week 3)
  The function in daily activities subscale of KOOS-12 will assess participants' ability to perform routine activities before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Babar Israr, MSPT, Principal Investigator — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar; Shakir Ullah, PhD, Study Director — Institute of Physical Medicine and Rehabilitation, Khyber Medical University Peshawar; Samra Farid, MSPT, Principal Investigator — Alkhidmat Hospital Peshawar
Locations (3):
- Pakistan (3):
  - Hayatabad Medical Complex Peshawar, Peshawar, KPK
  - Alkhidmat Hospital Peshawar, Peshawar, KPK
  - Bibi Zahida Memorial Hospital, NCS University System, Peshawar, KPK

IPD SHARING:
Plan to Share IPD: Yes
The study will make individual participant data (IPD) available to other researchers after the conclusion of the study. The IPD shared will include anonymized data related to the primary and secondary outcome measures, including depression scores, biochemical markers (e.g., TNF-α, IL-6, BDNF), EEG data, and other relevant clinical and demographic data collected during the trial. The data will be de-identified to ensure participant confidentiality. The data will be shared through an approved data repository or by direct request to the study's primary investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available 6 months after the study's completion and will remain accessible for a period of 5 years to facilitate further research.
Access Criteria: Access to the data will be granted to qualified researchers upon submission of a formal request that includes a research proposal outlining the intended use of the data. Requests will be reviewed by the study investigators and ethical review committee to ensure compliance with data privacy regulations.

REFERENCES:
- [Background] Farazdaghi M, Kordi Yoosefinejad A, Abdollahian N, Rahimi M, Motealleh A. Dry needling trigger points around knee and hip joints improves function in patients with mild to moderate knee osteoarthritis. J Bodyw Mov Ther. 2021 Jul;27:597-604. doi: 10.1016/j.jbmt.2021.04.011. Epub 2021 Apr 30. PMID 34391293
- [Background] Ceballos-Laita L, Jimenez-Del-Barrio S, Marin-Zurdo J, Moreno-Calvo A, Marin-Bone J, Albarova-Corral MI, Estebanez-de-Miguel E. Effects of dry needling on pain, pressure pain threshold and psychological distress in patients with mild to moderate hip osteoarthritis: Secondary analysis of a randomized controlled trial. Complement Ther Med. 2020 Jun;51:102443. doi: 10.1016/j.ctim.2020.102443. Epub 2020 May 18. PMID 32507443
- [Background] Ashraf F, Anwar K, Arshad H. Effects of muscle energy technique along conventional physical therapy after mesenchymal stem cell transplantation in knee osteoarthritis patients. Pak J Med Sci. 2024 Dec;40(11):2558-2564. doi: 10.12669/pjms.40.11.9605. PMID 39634887
- [Background] Goksen A, Can F, Yilmaz S, Korkusuz F. Comparison of different neuromuscular facilitation techniques and conventional physiotherapy in knee osteoarthritis. Turk J Med Sci. 2021 Dec 13;51(6):3089-3097. doi: 10.3906/sag-2101-298. PMID 34565133
- [Background] Sanchez-Romero EA, Pecos-Martin D, Calvo-Lobo C, Ochoa-Saez V, Burgos-Caballero V, Fernandez-Carnero J. Effects of dry needling in an exercise program for older adults with knee osteoarthritis: A pilot clinical trial. Medicine (Baltimore). 2018 Jun;97(26):e11255. doi: 10.1097/MD.0000000000011255. PMID 29952993